CLINICAL TRIAL: NCT03221491
Title: Comparison of Intravenous Patient-Controlled Analgesia With Different Background Infusion After Colorectal Surgery
Brief Title: Comparison of Patient-Controlled Analgesia With Different Background Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weifeng Tu (Other)
Responsible Party: Sponsor-Investigator, Weifeng Tu, Chief physician, Guangzhou General Hospital of Guangzhou Military Command
Organization: Guangzhou General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Different Background Infusion
Record Dates: First submitted 2017-07-16; First posted 2017-07-18 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Patient-Controlled Analgesia
Keywords: Analgesia; Colorectal Surgery; Background Infusion
MeSH Terms: conditions — Agnosia | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Background Infusion Group(Group B0) (Experimental): Patients in Group B0 receive analgesic regimens using Patient-Controlled Analgesia(PCA) with background infusion 0ml/h.
  Interventions: Device: Patient-Controlled Analgesia(PCA)
- Low Background Infusion Group(Group B1) (Experimental): Patients in Group B1 receive analgesic regimens using Patient-Controlled Analgesia(PCA) with background infusion 1ml/h.
  Interventions: Device: Patient-Controlled Analgesia(PCA)
- High Background Infusion Group(Group B2) (Experimental): Patients in Group B2 receive analgesic regimens using Patient-Controlled Analgesia(PCA) with background infusion 2ml/h.
  Interventions: Device: Patient-Controlled Analgesia(PCA)

INTERVENTIONS:
Device: Patient-Controlled Analgesia(PCA) — Patients receive analgesic regimens using Patient-Controlled Analgesia(PCA) with different background infusion.

SUMMARY:
In this study, the investigators investigated the efficacy, usefulness and analgesic consumption of three different patient-controlled analgesia(PCA) programmes:bolus dose alone without background infusion, bolus dose with low background infusion and bolus dose with high background infusion to evaluate postoperative analgesia for patients after laparoscopic colorectal surgery.

DETAILED DESCRIPTION:
There have been many studies using patient-controlled analgesia (PCA) and opioids for postoperative analgesia.Patient-controlled analgesia with opioids is now widely used after surgery for the treatment of acute postoperative pain. This technique provides effective pain treatment, adjusts the dose according to personal need and keeps plasma analgesic levels at a constant level,but the incidence of opioid-induced side-effects still be reported frequently.A proper PCA programme may increase efficiency of analgesic and decrease incidence of analgesic-induced side-effects.

In this study, 90 patients who is undergoing elective laparoscopic colorectal surgery will be randomly allocated into three groups (no background infusion group(Group B0),low background infusion group(Group B1) and high background infusion group(Group B2)). Patients in all groups will be given a patient-controlled analgesia (PCA) pump in post anesthetic recovery unit (PACU) after surgery.The PCA programme of Group B0 is dezocine 0.6mg/kg, flubiprofen 3mg/kg, diluted into 120ml and administer at a background infusion of 0ml/h, and a bolus of 4ml, with a lock-out of 15min. The PCA protocol of Group B1 is dezocine 0.6mg/kg,flubiprofen 3mg/k diluted into 120ml and administer at a background infusion of 1ml/h, and a bolus of 2ml, with a lock-out of 15min.The PCA protocol of Group B2 is dezocine 0.6mg/kg,flubiprofen 3mg/k diluted into 120ml and administer at a background infusion of 2ml/h, and a bolus of 2ml, with a lock-out of 15min.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists(ASA) Ⅰ-Ⅱ patient undergoing laparoscopic colorectal surgery
2. Written informed consent from the patient or the relatives of the participating patient.
3. BMI:18～30kg/m2

Exclusion Criteria:

1. Mental illness or cannot communicate.;
2. A second operation during the study;
3. Lung infection or sleep apnea syndrome;
4. Renal failure;
5. Alcohol or drug abuse;
6. Already taking gabapentin, pregabalin, benzodiazepin or antidepression drug;
7. Long-term use of analgesics,sedatives or non steroidal anti-inflammatory drugs history .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Dezocine consumption by patient-controlled analgesia | At 24 hours after surgery
  The total consumption of dezocine during 24 hours after surgery are recorded.

SECONDARY OUTCOMES:
The incidence rates of postoperative nausea and vomiting (PONV) | At 24 hours and 48 hours after surgery
  Measure whether nausea and vomiting exist and the level of severity.
Change in ramsay sedation score | At 0, 2, 4, 8, 24, 48 and 72 hours after surgery
  Measure sedation level by using ramsay sedation score.
Change in pain score | At 0, 2, 4, 8, 24, 48 and 72 hours after surgery
  Pain scores at rest and movement are evaluated with a numeric rating scale (NRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doyle E, Harper I, Morton NS. Patient-controlled analgesia with low dose background infusions after lower abdominal surgery in children. Br J Anaesth. 1993 Dec;71(6):818-22. doi: 10.1093/bja/71.6.818. PMID 8280546
- [Background] Yildiz K, Tercan E, Dogru K, Ozkan U, Boyaci A. Comparison of patient-controlled analgesia with and without a background infusion after appendicectomy in children. Paediatr Anaesth. 2003 Jun;13(5):427-31. doi: 10.1046/j.1460-9592.2003.01061.x. PMID 12791117
- [Background] White I, Ghinea R, Avital S, Chazan S, Dolkart O, Weinbroum AA. Morphine at "sub-analgesic" background infusion rate plus low-dose PCA bolus control pain better and is as safe as twice a bolus-only PCA regimen: a randomized, double blind study. Pharmacol Res. 2012 Aug;66(2):185-91. doi: 10.1016/j.phrs.2012.03.016. Epub 2012 Apr 6. PMID 22504462
- [Background] Hayes J, Dowling JJ, Peliowski A, Crawford MW, Johnston B. Patient-Controlled Analgesia Plus Background Opioid Infusion for Postoperative Pain in Children: A Systematic Review and Meta-Analysis of Randomized Trials. Anesth Analg. 2016 Oct;123(4):991-1003. doi: 10.1213/ANE.0000000000001244. PMID 27065359